CLINICAL TRIAL: NCT07221682
Title: Comparison For Ease Of Spinal Positioning & Duration Of Post-Op Analgesia Between Ultrasound Guided Supra-Inguinal Fascia Iliaca Block Vs Ultrasound Guided Infra-Inguinal Fascia Iliaca Block In Patients Undergoing Thigh & Knee Surgeries
Brief Title: Comparison of Supra vs Infra Inguinal Fascia Iliaca Blocks for Spinal Positioning and Analgesia in Lower Limb Surgery
Acronym: 27G
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Principal Investigator, Muhammad Shahid, Associate Professor, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202/IRB/SLMC/SWL
Record Dates: First submitted 2025-10-21; First posted 2025-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Post Operative Analgesia; Bradycardia; Hypotension Drug-Induced
Keywords: S-FICB; I-FICB; ASA; EOSP
MeSH Terms: conditions — Bradycardia; Hypotension

STUDY DESIGN:
Intervention Model Description: Group 1 will receive S-FICB and Group 2 will receive I-FICB
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP S-FICB (Other): Suprainguinal Facia Iliaca Block
  Interventions: Drug: USG GUIDED SUPRA-INGUINAL FASCIA ILIACA BLOCK
- GROUP I-FICB (Other): Infrainguinal Facia Iliaca Block
  Interventions: Drug: USG GUIDED INFRA-INGUINAL FASCIA ILIACA BLOCK

INTERVENTIONS:
Drug: USG GUIDED SUPRA-INGUINAL FASCIA ILIACA BLOCK — The S-FICB will be given as follows: With the patient in the proper position, the skin will be disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer will be moved laterally until the sartorius muscle is identified. The needle entry point will be anaesthetized with 2 ml 1% lidocaine and 23G spinal needle will be inserted. After negative aspiration, 1-2 mL of Inj Bupivacain 0.125% will be injected to confirm the proper injection plane between the fascia and the ilio-psoas muscle. A proper injection will result in the separation of the fascia iliaca by the local anesthetic in the medial-lateral direction from the point of injection as described. After the spread of the drug will be seen, the rest of the drug volume will be injected.
  Other Names: Sifi-B
  Arms: GROUP S-FICB
Drug: USG GUIDED INFRA-INGUINAL FASCIA ILIACA BLOCK — The I-FICB will be given in similar manner. In ultrasound guided I-FICB technique, a high frequency linear probe will be placed transversely at the level of the inguinal crease. After the femoral artery is identified, the probe will be moved laterally, and the hypoechoic iliopsoas muscle will be identified which is covered by the hyperechoic fascia iliaca. This fascia invests the femoral nerve medially and laterally covers the sartorius muscle. A needle will be inserted in-plane from lateral to medial and pierces the fascia iliaca at the junction of medial border of sartorius and iliopsoas muscle. Then Inj Bupivacain 0.125% will be deposited deep to fascia iliaca and will be seen spreading toward the femoral nerve medially.
  Other Names: Iifi-B
  Arms: GROUP I-FICB

SUMMARY:
Severe pain associated with thigh and knee fractures makes the positioning for regional anesthesia a challenge. Different modalities to make patient pain free for spinal positioning, post op analgesia and patient satisfaction including supra-inguinal fascia iliaca block (S-FIB) and infra-inguinal fascia iliaca blocks (I-FIB) have been studies. The aim of this study is to compare two blocks in patients undergoing thigh and knee surgeries.

A randomized controlled trial study design will be used and 60 patients fulfilling the inclusion criteria will be included. The patients will be divided into 2 groups by simple random sampling. Group A (S-FIB) (n = 30, those who will receive 30 ml of 0.125% bupivacaine) and Group B (I-FIB) (n = 30, those who will receive 30 ml of 0.125% bupivacaine). Depending on the allotted group, patients will be given the block under the guidance of ultrasound in the preoperative area. After block patients will be assessed for ease of spinal positioning using EOSP Scale, postoperative duration of analgesia and patient satisfaction using Likert Scale and data will be recorded on prescribed proforma.

All the findings will be noted in a specially designed proforma by the researcher. All the data collected will be entered and analyzed. Quantitative variables will be presented with mean ± SD. Independent sample t-test for duration of postoperative analgesia. Qualitative variables such as ease of spinal positioning and gender will be presented with Chi-Square. A p-value equal to or less than 0.05 will be considered significant.

DETAILED DESCRIPTION:
Patients fulfilling the inclusion criteria will be included. Patients will be optimized for dressing. A detailed history will be taken regarding the mode of injury, any pre-existing disease and previous surgery followed by the local examination of the patient will be done to rule out any systemic disease. Informed consent will be taken. These patients will be divided into 2 groups by Computer-generated random numbers and group assignment will be done by sequentially numbered opaque envelopes. The envelope will be opened just before the procedure by the anaesthesiologist performing the block. The observer (another anaesthesiologist) and patients will be unaware of the group and procedure performed. Group A (Supra-inguinal Fascia Iliaca Block) and Group B (Infra-inguinal Fascia Iliaca Block). The monitors of electrocardiogram, pulse oximetry and non-invasive blood pressure in induction room will be connected. For drug and fluid administration, an intravenous cannula of suitable size will be obtained. Pre-procedural pain will be assessed during rest as well as on movement (15° passive elevation) of the affected limb and will be recorded on numeric pain rating scale (NRS) [0 = no pain; 10 = worst imaginable pain]. The blocks will be performed in supine position and strict sterile technique will be followed. Both the blocks will be performed as per the standard technique. The site to be blocked will be painted with 5% povidone-iodine followed by spirit and will be draped. A linear 7-13 mhz ultrasonography probe (sonoscape S 11plus, digital colour doppler ultrasound., Guangdong, China) will be used with in-plane approach of needle. Group A (S-FIB) (n = 30, those who will receive a S-FIB with 30 ml of 0.125% bupivacaine) and group B (I-FIB) (n = 30, those who will receive a I-FIB with 30 ml of 0.125% bupivacaine). Depending on the allotted group, patients will be given the block under the guidance of ultrasound in the preoperative area by an experienced anesthesiologist with more than two years' experience. The S-FIB will be given as follows: With the patient in the proper position, the skin will be disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer will be moved laterally until the sartorius muscle is identified. The needle entry point will be anaesthetized with 2 ml 1% lidocaine and 23G spinal needle will be inserted. After negative aspiration, 1-2 ml of Inj Bupivacain 0.125% will be injected to confirm the proper injection plane between the fascia and the ilio-psoas muscle. A proper injection will result in the separation of the fascia iliaca by the local anesthetic in the medial-lateral direction from the point of injection as described. After the spread of the drug will be seen, the rest of the drug volume will be injected.

The I-FIB will be given in similar manner. In ultrasound guided I-FIB technique, a high frequency linear probe will be placed transversely at the level of the inguinal crease. After the femoral artery is identified, the probe will be moved laterally, and the hypoechoic iliopsoas muscle will be identified which is covered by the hyperechoic fascia iliaca. This fascia invests the femoral nerve medially and laterally covers the sartorius muscle. A needle will be inserted in-plane from lateral to medial and pierces the fascia iliaca at the junction of medial border of sartorius and iliopsoas muscle. Then Inj Bupivacain 0.125% will be deposited deep to fascia iliaca and will be seen spreading toward the femoral nerve medially.

A numerical rating scale (NRS) pain score will be recorded after the block. The onset time to achieve NRS pain score of 4 or less than 4 will be noted on prescribed proforma for both groups. The patients will be made to sit for spinal anesthesia and ease of spinal positioning according to the scale (0,1,2,3) , will be noted after preloading with ringer lactate solution @80ml/kg. The spinal anaesthesia will be performed using 27G spinal needle (Quincke) with 0.75% bupivacaine solution (2ml) in both groups. The monitors of electrocardiogram, pulse oximetry, non-invasive blood pressure and urine output will be monitored according to ASA standard. After completion of surgery patient will be shifted to respective ward where trained doctor and staff will monitor the patient. The NRS score will be measured immediately postoperatively and at intervals of 2 hours for a period of 12 hours. If the NRS score will be >4, rescue analgesia will be given; an injection of paracetamol 15 mg/kg will be given over a period of 10 to 15 minutes as an intravenous infusion. Inj nalbuphine 0.1mg/kg will be given for breakthrough pain. Total dose of intravenous nalbuphine will be recorded in 1st 12hrs. Patient satisfaction will be measured on a 1-5 Likert Scale after 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Both Genders (Male /Female).
2. Age between 30 years to 60 years.
3. ASA Class I, II, III.

Exclusion Criteria:

1. Patient refusal
2. Other distracting painful pathology
3. Any contraindication to Spinal Anesthesia or peripheral nerve blocks
4. Coagulopathic disorders
5. Patients with significant cognitive impairment
6. Patients with no pain while sitting by themselves without any support
7. H/O polytrauma involving other limbs
8. H/O allergy to the drugs used in study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Ease of Spinal Positioning | From performance of block to spinal anesthesia procedure begins
  The ease of spinal positioning (EOSP) will be assessed on the scale of 0-3 0= unable to position
  1. patient had abnormal posturing due to pain and required support for positioning
  2. mild discomfort but does not require support for positioning
  3. optimal condition where the patient was able to position himself without pain

SECONDARY OUTCOMES:
Post Op Analgesia | From Performance of Block to First Rescue Analgesia e.g. at 0,2,4,6 upto 12 hours
  Duration of Post Op Analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- Sahiwal Medical College Sahwal, Sāhīwāl, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request after completion of study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: November 2025
Access Criteria: On Demand